CLINICAL TRIAL: NCT02765893
Title: Indwelling vs Immediate Removal of Foley Catheter After Robotic Assisted Laparoscopic Sacrocolpopexy: a Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantic Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 791664-1
Record Dates: First submitted 2016-05-05; First posted 2016-05-09 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Urinary Retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Foley (No Intervention): Patients will have Foley in place overnight after completion of surgery, which is currently standard of care at our institution.
- No Foley (Active Comparator): Patients will have Foley catheter removed 6 hours post-op.
  Interventions: Other: No Foley

INTERVENTIONS:
Other: No Foley — Patients will have Foley catheter removed 6 hours post-op.
  Arms: No Foley

SUMMARY:
This is a prospective, comparative randomized study. Our study population includes women with pelvic organ prolapse undergoing a robotic assisted laparoscopic sacrocolpopexy.

The two groups will include the study group, who will have their Foley catheter removed 6 hours post-op, and the control group who will have an indwelling Foley catheter overnight. The two groups will be assigned according REDCap randomization system.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-75
* Pelvic organ prolapse requiring robotic assisted, laparoscopic sacrocolpopexy.

Exclusion Criteria:

* Intraoperative complications necessitating a post-operative Foley

  * Cystotomy
  * EBL >500mL
  * Bowl injury
* Pre-operative urinary retention requiring an indwelling catheter

Ages: 19 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-12; Primary Completion 2017-09-21 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
Urinary retention | 6 hours after discharge from PACU
  Patients in the intervention group will have their Foley catheter removed up to 6 hours after discharge from the PCA. They will then have to undergo a voiding trial

SECONDARY OUTCOMES:
Urinary Tract Infections | 30 day post op
  All UTIs will be documented up to 30days post op.
Post-operative complications | 30 days post op
  Post-operative complications

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantic Health, Morristown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geller EJ, Siddiqui NY, Wu JM, Visco AG. Short-term outcomes of robotic sacrocolpopexy compared with abdominal sacrocolpopexy. Obstet Gynecol. 2008 Dec;112(6):1201-1206. doi: 10.1097/AOG.0b013e31818ce394. PMID 19037026
- [Background] Siddiqui NY, Geller EJ, Visco AG. Symptomatic and anatomic 1-year outcomes after robotic and abdominal sacrocolpopexy. Am J Obstet Gynecol. 2012 May;206(5):435.e1-5. doi: 10.1016/j.ajog.2012.01.035. Epub 2012 Feb 1. PMID 22397900
- [Background] Alessandri F, Mistrangelo E, Lijoi D, Ferrero S, Ragni N. A prospective, randomized trial comparing immediate versus delayed catheter removal following hysterectomy. Acta Obstet Gynecol Scand. 2006;85(6):716-20. doi: 10.1080/00016340600606976. PMID 16752265
- [Background] Ahmed MR, Sayed Ahmed WA, Atwa KA, Metwally L. Timing of urinary catheter removal after uncomplicated total abdominal hysterectomy: a prospective randomized trial. Eur J Obstet Gynecol Reprod Biol. 2014 May;176:60-3. doi: 10.1016/j.ejogrb.2014.02.038. Epub 2014 Mar 4. PMID 24670774
- [Background] Zhang P, Hu WL, Cheng B, Cheng L, Xiong XK, Zeng YJ. A systematic review and meta-analysis comparing immediate and delayed catheter removal following uncomplicated hysterectomy. Int Urogynecol J. 2015 May;26(5):665-74. doi: 10.1007/s00192-014-2561-0. Epub 2014 Nov 15. PMID 25398392
- [Background] Summitt RL Jr, Stovall TG, Bran DF. Prospective comparison of indwelling bladder catheter drainage versus no catheter after vaginal hysterectomy. Am J Obstet Gynecol. 1994 Jun;170(6):1815-8; discussion 1818-21. doi: 10.1016/s0002-9378(94)70358-2. PMID 8203443
- [Background] Dobbs SP, Jackson SR, Wilson AM, Maplethorpe RP, Hammond RH. A prospective, randomized trial comparing continuous bladder drainage with catheterization at abdominal hysterectomy. Br J Urol. 1997 Oct;80(4):554-6. doi: 10.1046/j.1464-410x.1997.t01-1-00376.x. PMID 9352691
- [Background] Dunn TS, Shlay J, Forshner D. Are in-dwelling catheters necessary for 24 hours after hysterectomy? Am J Obstet Gynecol. 2003 Aug;189(2):435-7. doi: 10.1067/s0002-9378(03)00496-4. PMID 14520213
- [Derived] Ellahi A, Stewart F, Kidd EA, Griffiths R, Fernandez R, Omar MI. Strategies for the removal of short-term indwelling urethral catheters in adults. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD004011. doi: 10.1002/14651858.CD004011.pub4. PMID 34184246